Protocol No.: 201205030RIB Confidential

## **CLINICAL STUDY PROTOCOL**

## Screening for Colorectal Neoplasms with the Fecal Testing: a Population-based Randomized Study

Protocol Number: 201205030RIB

ClinicalTrial.gov Number: NCT 01741363

Indication: Colorectal Neoplasms
Principal Investigator: Han-Mo Chiu, M.D., Ph.D.

Version Number: V1.0

Date May-30-2012

Funding Support: Health Promotion Administration, Ministry of Health

and Welfare

All the information disclosed or provided by the Health Promotion Administration, Ministry of Health and Welfare or produced during the clinical trial, including this protocol, the CRFs, the Investigator Brochure, and the results obtained during the clinical trial, is confidential and is intended for the use of clinical investigators, and any person under his/her authority agree to keep confidential.

Protocol version: V1.0 Date: May-30-2012

Protocol No: 201205030RIB

Confidential

ABSTRACT

Screening for stomach diseases and colorectal neoplasms with

the fecal testing: a population-based randomized study

Growing body of evidences have shown that fecal immune test (FIT)

outperform guaiac fecal occult blood test (gFOBT) in terms of sensitivity,

neoplasm detection rate and public participation. Though direct outcome

evidence is still lacking for FIT, it is anticipated to have higher colorectal cancer

(CRC) mortality and incidence reduction compared with gFOBT. In Taiwan,

nation-wide CRC screening program has been launched since the year of

2004 ,which provides biennial FIT screening for adults aged 50 to 75 years.

Currently available data from the Bureau of Health Promotion has shown a

significant stage-shift effect, an early indicator of screening effectiveness, by this

screening program.

Nevertheless the aforementioned advantages of FIT, missed neoplasms and

interval cancer still exists under the current one-day stool sampling method

with biennial screening interval, which might affect the effectiveness of overall

screening program. Increase the number of stool samples or shortening of

screening interval may be helpful for early detection of clinically significant

neoplasms but it remains unclear whether such an approach may lower the

screenee compliance or public participation. Moreover, its impact on the

demand of confirmatory colonoscopy and cost-effectiveness of the whole

screening program is still largely unknown and need to be further investigated.

In this study, we aim to randomly allocate screening attendee to one of the

Protocol version V1.0 Data:May-30-2012

Protocol No: 201205030RIB

Confidential

following four arms: one-day sampling with annual screening, one-day sampling

with biennial screening, two-day sampling with annual screening, and two-day

sampling with biennial screening. Participation rate, positive rates of FIT,

detection rate for neoplasms, positive predictive value, and long-term outcome

including cancer incidence and mortality will be calculated and compared among

four groups. In addition, cost-effectiveness analysis will be also conducted using

previously established Markov model of CRC natural history using the results

ascertained from this trial.

The abundant results from this trial will be helpful for assessing the feasibility

of increasing stool sampling and shortening screening interval in population

setting, their long-term effects, and cost-effectiveness.

However, in Taiwan, although the incidence of colorectal cancer is rapidly

increasing, *Helicobacter pylori*-related upper GI pathologies remain highly

prevalent, which may imply that mass screening solely based on FIT could be

insufficient as significant upper GI pathologies can be missed. Since FIT dose not

predict upper GI pathologies, the adjuncts of *H. pylori* stool-antigen test (HpSA)

may be a potential candidate to realize a pan-detecting assay based on stool

samples in a population in which both lower and upper GI lesions are equally

prevalent.

Protocol version V1.0 Data:May-30-2012